CLINICAL TRIAL: NCT03144102
Title: The Effects of Combining Transcranial Direct Current Stimulation (tDCS) With VR-based Motor Training in Hemiparetic Stroke Patients
Brief Title: Combining tDCS With VR-based Motor Training in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Neuroelectrics Corporation (Industry)
Responsible Party: Principal Investigator, Paul Verschure, Prof., Universitat Pompeu Fabra
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCSRGS
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Virtual Reality Based Therapy; Anodal tDCS; Occupational Therapy; Sham tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- VR-based motor rehabilitation with tDCS (Experimental)
  Interventions: Behavioral: Virtual Reality-based therapy for upper-limbs motor rehabilitation; Device: Anodal transcranial direct-current stimulation (tDCS)
- Occupational Therapy with tDCS (Active Comparator)
  Interventions: Device: Anodal transcranial direct-current stimulation (tDCS); Behavioral: Occupational Therapy for upper-limbs motor rehabilitation
- VR-based motor rehabilitation with sham tDCS (Sham Comparator)
  Interventions: Behavioral: Virtual Reality-based therapy for upper-limbs motor rehabilitation; Device: Sham transcranial direct-current stimulation (tDCS)
- Occupational Therapy with sham tDCS (Sham Comparator)
  Interventions: Behavioral: Occupational Therapy for upper-limbs motor rehabilitation; Device: Sham transcranial direct-current stimulation (tDCS)

INTERVENTIONS:
Behavioral: Virtual Reality-based therapy for upper-limbs motor rehabilitation — During each session, the subject will perform 4 VR-based exercises that involve reaching, grasping, and intercepting virtual objects. The training will last a total of 30 min per session.
  Arms: VR-based motor rehabilitation with sham tDCS; VR-based motor rehabilitation with tDCS
Device: Anodal transcranial direct-current stimulation (tDCS) — Concurrent anodal tDCS on sensorimotor cortex on the ipsilesional hemisphere.
  Arms: Occupational Therapy with tDCS; VR-based motor rehabilitation with tDCS
Behavioral: Occupational Therapy for upper-limbs motor rehabilitation — During each session, the subject will perform 4 occupational therapy exercises that involve reaching, grasping, and intercepting objects. The training will last a total of 30 min per session.
  Arms: Occupational Therapy with sham tDCS; Occupational Therapy with tDCS
Device: Sham transcranial direct-current stimulation (tDCS) — Concurrent sham tDCS on sensorimotor cortex on the ipsilesional hemisphere.
  Arms: Occupational Therapy with sham tDCS; VR-based motor rehabilitation with sham tDCS

SUMMARY:
Stroke represents one of the main causes of adult disability and will be one of the main contributors to the burden of disease in 2030. However, our healthcare systems do not have enough resources to cover the current demand let alone its future increase. There is a need to deploy new approaches that advance the current rehabilitation methods and enhance their efficiency.

One of the latest approaches used for the rehabilitation of a wide range of deficits of the nervous system is based on virtual reality (VR) applications, which combine training scenarios with dedicated interface devices. On the other hand, recent studies have shown the potential of transcranial direct current stimulation (tDCS) to restore motor function in hemiparetic stroke patients. It must be emphasized, however, that so far little work exists on the quantitative assessment of the clinical impact of VR based approaches in combination with tDCS protocols. We hypothesize that the combination of VR-based motor rehabilitation protocols with concurrent anodal tDCS can boost functional recovery, and may achieve superior effects when compared to 3 alternative treatments: 1) VR without tDCS, 2) occupational therapy with tDCS, and 3) occupational therapy without tDCS.

The findings derived from this study will contribute to establish a novel and superior neurorehabilitation paradigm that can accelerates the recovery of hemiparetic stroke patients. Besides the clinical impact, such achievement could have relevant socioeconomic impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiparesis secondary to first ever ischemic or hemorrhagic stroke (Medical Research Council score > 2).
* Older than 18 years old.
* Sufficient cognitive capacity to understand and follow the experimental instructions (Mini-Mental State Evaluation > 20).

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Epilepsia and metal implants. A diagnostic EEG will be performed by the Department of Clinical Neurophysiology of the hospital to detect epileptic paroxysmal in order to include or exclude patients in the study.
* Low Cognitive capabilities that prohibits the execution of the experiment Arteriovenous malformation
* Severe associated impairment such as spasticity, communication disabilities (sensorial, mixed or global aphasia or apraxia), major pain or other neuromuscular impairments or orthopaedic devices that would interfere with the correct execution of the experiment (Modified Ashworth Scale > 3)
* History of serious mental-health problems in acute or sub acute phase
* Refusal to sign the consent form
* Previous surgeries opening the skull.
* Active or recent substance abuse or dependence within the past year.
* Pregnancy, breastfeeding, unwillingness to practice birth control during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-12-08 (Estimated); Study Completion 2021-06-08 (Estimated)

PRIMARY OUTCOMES:
Change of arm/hand function as captured by the upper extremity Fugl-Meyer assessment scale | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)

SECONDARY OUTCOMES:
Change of Independence as captured by Barthel scale | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)
Change of motor function in ADLs as captured by Chedoke Arm and Hand Activity Inventory (CAHAI) scale | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)
Change of interhemispheric balance as captured by EEG recordings | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)
Change of spasticity in proximal and distal muscles as captured by Ashworth scale | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)
Change of spatial hemineglect as captured by the Star cancellation test | At baseline, at 2-weeks (after intervention), and at 8-weeks (follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- Unitat de Rehabilitació de l'Hospital Vall d'Hebron, Barcelona, Spain